CLINICAL TRIAL: NCT01953718
Title: A Retrospective Study of the Effects of Different Parameters on Motor Symptoms of PD in Bilateral STN Stimulation
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Chen Ling, MD,PhD, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: [2008]20; 10151008901000187 (Other Grant/Funding Number: GNSF)
Record Dates: First submitted 2013-09-26; First posted 2013-10-01 (Estimated); Last update posted 2013-10-10 (Estimated); Status verified 2013-10

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
The purpose of this study is to assess the impact of different parameters (voltage, pulse width, frequency) of subthalamic nucleus (STN) deep brain stimulation (DBS) on motor symptoms in patients with Parkinson's disease (PD).

DETAILED DESCRIPTION:
In this observational study, we will retrospectively analyze the one-year follow-up data of 27 PD patients who received bilateral STN DBS in the First Affiliated Hospital of Sun Yat-sen University in the years 2008-2012. The data, including parameter settings and severity of motor symptoms indicated by Unified Parkinson's Disease Rating Scale (UPDRS) Part III scores, was collected during the patients' annual visit to the hospital for reprogramming. A correlation analysis will be conducted to investigate the relationship between change of a specific parameter and the subsequent change of motor scores.

ELIGIBILITY:
Inclusion Criteria:

* PD patients treated with bilateral STN DBS in the First Affiliated Hospital in the years 2008-2012

Exclusion Criteria:

* Simultaneous participation in another clinical trial
* Dementia (Mini Mental State Examination < 26)
* Removal of DBS electrodes
* Loss to follow-up

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PD patients who received bilateral STN DBS in the First Affiliated Hospital of Sun Yat-sen University
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2013-07; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change of parameters (voltage, pulse width, frequency) during follow-up | at 12 months
Change of UPDRS Part III score and the relation to parameters | at 12 months
Changes of tremor, rigidity, bradykinesia and postural stability scores evaluated by UPDRS Part III and the relation to parameters | at 12 months

SECONDARY OUTCOMES:
Change of daily levodopa equivalent dosage (LED) during follow-up | at 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong, China